CLINICAL TRIAL: NCT03068013
Title: Effectiveness of a Brief Manualized Intervention Managing Cancer and Living Meaningfully (CALM) Adapted to the Italian Cancer Care Setting. Study Protocol for a Randomized Controlled Trial
Brief Title: Managing Cancer and Living Meaningfully (CALM) Adapted to Italian Cancer Care Setting
Acronym: CALM-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Luigi Grassi, Professor and Chair of Psychiatry, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAR-2015
Record Dates: First submitted 2016-09-24; First posted 2017-03-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Quality of Life
Keywords: CALM; Depression; Demoralization; Cancer; Spirituality; Psychotherapy; Quality of Life; Anxiety; Post-Traumatic Growth
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Cancer Living Meaningfully (Experimental): Patients in the experimental group will receive the brief, individual, manualized CALM intervention, a semi-structured psychotherapy designed for patients with advanced cancer. CALM was developed based on empirical results, clinical observation and the theoretical foundations of supportive-expressive and existential approaches, as well psychodynamic and attachment theories. The sessions are delivered bimonthly over a period of 6 months. Sessions are reviewed to ensure treatment fidelity.
  Interventions: Behavioral: CALM
- Supportive psycho-oncology intervention (Active Comparator): Supportive psycho-oncology intervention (SPI) includes counseling, psychoeducation and crisis intervention, which is the usual care intervention provided in our centres.
  Interventions: Behavioral: SPI

INTERVENTIONS:
Behavioral: CALM — CALM intervention covers four domains, namely: 1) Symptom management and communication with health care providers; 2) Changes in self and relations with close others, 3) Spiritual well-being, sense of meaning and purpose, 4) Preparing for the future, sustaining hope and facing mortality
  Arms: Managing Cancer Living Meaningfully
Behavioral: SPI — Active Comparator: Supportive psycho-oncology intervention Supportive psycho-oncology intervention (SPI) includes counseling, psychoeducation and crisis intervention, which is the usual care intervention provided in our centres.
  Arms: Supportive psycho-oncology intervention

SUMMARY:
Background: Patients with advanced cancer suffer from a variety of psycho-social symptoms that impair quality of life and may benefit from psychotherapeutic treatment. We describe here the methodology of a randomized controlled trial to test the effectiveness of a novel and brief semi-structured psychotherapeutic intervention, called Managing Cancer and Living Meaningfully (CALM), originally developed in Canada and now cross-culturally tested in Italy.

Methods/Design: The study is a single-blinded randomized controlled trial with 2 conditions: CALM intervention versus nonspecific supportive intervention (SPI) and assessments at baseline, 3 and 6 months. The coordinating site is the Program on Psycho-Oncology and Psychiatry in Palliative Care, University of Ferrara and Integrated Department of Mental Health, S. Anna University Hospital, in Ferrara, Italy. Another centre from northern and southern Italy will collaborate. Eligibility criteria include: ≥ 18 years of age; Italian fluency; no cognitive impairment; and diagnosis of advanced cancer. The intervention consists of 12 sessions , following the CALM manual and allowing for flexibility to meet individual patients' needs. It is delivered over a 6-month period and provides reflective space for patients (and their primary caregivers) to address 4 main domains: symptom management and communication with health care providers; changes in self and relations with close others; sense of meaning and purpose; and the future and mortality. The primary outcome is depression and the primary endpoint is at 6 months. Secondary outcomes include demoralization, generalized anxiety, death anxiety, spiritual well-being, quality of life, attachment security, posttraumatic growth, communication with partners, and satisfaction with clinical interactions.

Discussion: This trial is being conducted to determine the effectiveness of CALM in an Italian cancer setting. The intervention has potential cross-national relevance and, if shown to be effective, has the potential to be disseminated as a new approach in oncology to relieve distress and promote psychological well-being in patients with advanced cancer.

DETAILED DESCRIPTION:
The study is coordinated by the Program on Psycho-Oncology and Palliative Care, University of Ferrara Northern Italy. Another centre from northern Italy will collaborate. The study is designed as a single-blinded randomized-controlled trial with two arms. Participants in the experimental group will receive the CALM intervention, while those in Control Group will receive a supportive intervention, which is usual psycho-oncology care in our settings.The primary outcome is depression. The primary endpoint is 6 months. Secondary outcomes include demoralization, generalized anxiety, death anxiety, spiritual well-being, quality of life, attachment security, posttraumatic growth, communication with partners, and satisfaction with clinical interactions.The study has received approval from Ethical Committees.

Interventions:Patients in the experimental group will receive the CALM intervention, a semi-structured psychotherapy designed for patients with advanced cancer. In this Italian adaptation, CALM consists of 12 individual sessions (45-60 minutes each), instead of the original 6 sessions. The sessions are delivered bimonthly over a period of 6 months.

The intervention covers four domains: 1) Symptom management and communication with health care providers; 2) Changes in self and relations with close others; 3) Spiritual well-being, sense of meaning and purpose; 4) Preparing for the future, sustaining hope and facing mortality.

Non-manualized supportive psycho-oncology intervention (SPI):The Control group intervention includes counseling, information, crisis intervention, which is the usual care intervention provided in our center. As with CALM patients, SPI patients receive up to twelve sessions of individual therapy during a period of 6 months.

Inclusion criteria are:18 years of age or more;fluency in Italian language; absence of cognitive deficit documented in the clinical records;diagnosis of "wet" stage IIIB or IV lung cancer; any stage of pancreatic cancer, stage III or IV ovarian and fallopian tube cancers, or other stage IV gynecological cancer; and stage IV breast, genitourinary, gastrointestinal, melanoma, sarcoma, or endocrine cancers (all with an expected survival of 12-18 months); a score ≥10 at the Patient Health Questionnaire and/or ≥ 20 at the Death and Dying Distress Scale. Exclusion criteria are: language barriers hindering psychotherapy;inability to commit to the required 12 sessions; concomitant psychotherapy.

Randomization procedure:Study participants are randomly assigned to receive either CALM or SPI. After obtaining informed consent , a research assistant includes patient's data on the random allocation list and informs the PI's about treatment allocation (CALM or SPI). The patient is not informed about treatment condition (CaLM or SPI).

Measures:The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression. It is composed by nine items, reflecting DSM-IV criteria for major depression. A four-point Likert scale scores from 0 (not at all) to 3 (nearly every day), with a cut-off score of ≥10 suggesting depression. For study purposes, two additional items assessing self-harm intention and rating how difficult these symptoms have made it to do lead one's life, have been included.The Demoralization Scale (DS) is a 24-item self-report tool assessing demoralization components of loss of meaning and purpose, dysphoria, disheartenment and helplessness. Items are scored on a five-point Likert scale ranging from 0 (never) to 4 (all the time). Low levels of demoralization were indicated by a score 10, moderate demoralization by a score 11-36, and high demoralization by a score > 37.The Generalized Anxiety Disorder Questionnaire (GAD-7) is a 7-item self-report instrument screening the severity of GAD symptoms. Items are scored on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). Scores ≤4 indicate absence of anxiety, scores from 5 to 9 suggest that mild anxiety is present, and scores from 10 to 15 indicate moderate levels of anxiety. An eighth item rating how difficult these symptoms have made it to lead one's daily life has been included. The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-SP)[v] is a 12-item self-report tool, exploring spiritual well-being, in terms of sense of meaning, faith and inner peace. Items are scored on a five-point Likert scale from 0 (not at all) to 4 (very much), with higher scores indicating a greater spiritual wellbeing.The Posttraumatic Growth Inventory (PTGI) is a 21-item self-report measure of positive psychological changes after traumatic events. It consists of four subscales: New Possibilities, Appreciation of Life, Relating to Others and Spiritual Change. Items are scored on a three-point Likert scale ranging from 0 (not at all) to 2 (very much) with higher scores indicating greater post-traumatic growth.The Quality of Life at the End of Life-Cancer Scale (QUAL-EC) is a self- report measure of quality of life in patients near the end of life. It originally consists of four subscales: Symptom Control, Relationship with Health Care Providers, Preparation for End of Life and Life Completion. For this study purposes, the symptom control subscale is not included, thus only items 4-17 are used. Items are scored on a five-point Likert scale ranging from 1 (not at all) to 5 (completely), with higher scores indicating higher quality of life.The Death and Dying Distress Scale (DADDS), is a 15-item self-report measure assessing specific concerns of advanced cancer patients about end of life, feeling a burden to others and wasted opportunities. It is scored on a six-point Likert scale from 0 (no distress) to 5 (very much distress), with higher scores indicating higher death anxiety and distress.The Experiences in Close Relationships Inventory Modified Short Form Version (ECR-M16), is used in its 16-item self-report form to measure the attachment style. The scale yields scores on two dimensions of attachment: avoidance and anxiety. Items are scored on a seven-point Likert scale ranging from 1 (disagree) to 7 (agree), with a total sum score on each subscale ranging from 16 to 56. Higher scores on both subscales indicate higher attachment insecurity.The Memorial Symptom Assessment Scale (MSAS) [x]assesses the disease symptom severity. The scale, in its shortened version (MSAS- short form), measures the presence and severity of 28 common physical symptoms of cancer. Items are scored on a five-point Likert scale ranging from 0 (not at all) to 4 (very much).

The Couple Communication Scale (CCS) is used for participants who have a partner. The 10-item CCS taken from the PREPARE/ENRICH Inventory is concerned with an individual's feelings, beliefs, and attitudes about the communication in his/her romantic relationship. Each item is scored from 1 (strongly disagree) to 5 (strongly agree).

Intervention and control participants will complete the Clinical Evaluation Questionnaire (CEQ) at 3 and 6-months. The CEQ is a seven-item self-report questionnaire which assesses the amount of clinical benefit patients have experienced by from therapy at the time of the assessment. Items are rated from 0 to 4, with 0 (no clinical benefit) and 4 (a great clinical benefit).Satisfaction of patients will also be qualitatively assessed by inviting them to share comments in a written form after completing CEQ questionnaire.

Assessment:At baseline (T0), participants provide demographics and medical and treatment data using a standardized questionnaire and will complete all outcome measures, with the exception of the CEQ. The PHQ-9 and DADDS are first administered to assess eligibility prior to study entry, followed by the remaining baseline outcomes. Follow-up assessments on all outcomes are collected at three months (T1) and six months (T2). The CEQ is administered only at three months (T1) and six months (T2) as it is an evaluation of the intervention received to date. At T2, participants will also be queried about their having remained blind (or not) to randomization.

Statistical methods:To calculate the required sample size, we used a validated, manualized online power and sample size calculator that is ideal for longitudinal multilevel designs, GLIMMPSE [ ]. A total sample size estimate for our primary hypothesis, that the treatment group (CALM) will demonstrate a greater higher improvement ind depressive symptoms (PHQ-9) at follow-up periods, as compared to the control group (SPI), was derived with a target power of 80% and alpha of .05 and with estimated mean scores, with variability, and cross-time correlations entered. For the primary hypothesis, the calculated total sample size is 124 patients (62 patients per treatment arm). To account for anticipated attrition while maintaining the targeted power, we used the following equation to calculated an adjusted sample size: N = N0 * (1 + DRP), where N0 = original estimated sample size required at baseline; DRP = anticipated dropout rate across participants. For an anticipated completion rate of 70% rate (30% dropout rate), the adjusted sample size for this attrition rate is N = 124 * (1 + .30) = 161.2. The adjusted sample size at baseline will therefore be 162, with 81 patients per treatment arm.

Statistical analyses will be carried out by using SPSS Statistics program. For the final analyses we will use an intention-to-treat approach (ITT) and compare patients in the assigned treatment arms. To test the pPrimary hypothesis : we hypothesize that mean depression scores in the intervention arm will be lower than in the control arm at 3 and 6 months, . We will use multilevel modeling (MLM) with maximum likelihood estimation to conduct the intent-to-treat analysis in testing hypotheses. MLM includes all participants, including those with missing data, in model estimation and also accounts for both inter-center and intra-center variability.To test for treatment-arm differences, we will compare the CALM and SPI groups on the primary outcome of PHQ-9 scores and on the secondary outcomes at the follow-up periods. This will entail the following set of MLM analyses:i)We will first test the level-1 predictor of Time, coded for the primary hypothesis as a categorical variable representing baseline and the 6-month follow-up period (primary endpoint). To code time for tests of secondary hypotheses, the categorical time variable will include baseline and the 3-month (secondary endpoint) and 6-month follow-up periods. ii)Next, we will add the level-2 treatment-group main effect and the cross-level treatment group x time interactions to test the hypothesized treatment-group differences at follow-up periods. Pairwise comparisons will evaluate the treatment-group difference at each follow-up period.iii)We will finally test whether the fixed effects in step ii change when any identified covariates are added to control for their effects. As a sensitivity analysis, we will use multiple imputation to examine the influence of missing values. Lastly, prior trial results suggest that there may be arm differences in the processing of death-related distress such that individuals with moderate death anxiety tend to be more responsive to the intervention than either those with low death anxiety (approximately the lower third of the distribution) or those with high death anxiety (the upper third). We will conduct a sub-analysis to confirm this effect, by examining the effect of removing individuals with low and high death anxiety scores at baseline (i.e., DADDS < 15), following the Canadian protocol.

We will also qualitatively analyze the participants' comments about CALM and SPI on the CEQ. NVivo Plus software package will be used for the qualitative analysis of data.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or more
2. fluency in Italian language;
3. no cognitive impairment;
4. confirmed or working diagnosis of "wet" stage IIIB (those not treated with curative intent) or IV lung cancer; any stage of pancreatic or stage IV GI cancer, stage III or IV ovarian and fallopian tube cancers, or other stage IV gynecological cancer; and stage IV breast, genitourinary, sarcoma, melanoma or endocrine cancers (expected survival of 12-18 months); a score ≥10 at the Patient Health Questionnaire (PHQ9) or ≥ 20 at the Death and Dying Distress Scale (DDAS). -

Exclusion Criteria:

1. communication difficulties;
2. inability to commit to the required 6 sessions (i.e., too ill to participate, lack of transportation, etc.);
3. actively seeing a psychotherapist, and

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PHQ - depression | Changes in depression levels by PHQ will be assessed at baseline to assess eligibility, after 3 months and after 6 months
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression. It is composed by nine items, reflecting Diagnostic and Statistical Manual-IV criteria for major depression. A four-point Likert scale scores from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. A cut-off point of ≥10 is used as recommended for the screening of depression,but further analysis will be done according to other cut-off scores recommended to classify the type of depression, specifically, no depression/minimal (score 0-4), mild depression (score 5-9), moderate depression (score10-14), moderately severe depression (score 15-19), severe depression (score 20-27). For study purposes, two additional items assessing intent to cause self-harm and rating how difficult these symptoms have made it to do work, take care of things at home, or get along with other people, have been included.

SECONDARY OUTCOMES:
Generalized anxiety levels measured by GAD 7-generalized anxiety | Baseline, after 3 months and after 6 months
  The Generalized Anxiety Disorder Questionnaire (GAD-7)is a 7-item self-report measure designed to screen the severity of GAD symptoms. Items are scored on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day) with a total score ranging from 0 to 21. Scores up to 4 indicate absence of anxiety, scores from 5 to 9 indicate the presence of mild anxiety, scores from 10 to 15 indicate moderate anxiety. An eighth item rating how difficult these symptoms have made it to do work, take care of choirs at home, or get along with other people, has been included.
Death and dying distress measured DADDS-Death and dying distress scale | Baseline, after 3 months and after 6 months
  The Death and Dying Distress Scale (DADDS) is a 15-item self-report measure assessing specific concerns of advanced cancer patients about end of life, feeling a burden to others and wasted opportunities. It is scored on a six-point Likert scale from 0 (no distress) to 5 (very much distress), with a total score ranging from 0 to 75, a greater score indicating higher death anxiety and distress.
Spiritual well being, measured by FACIT-Sp - Spiritual well-being | Baseline, after 3 months and after 6 months
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-SP) is a 12-item self-report measure of spiritual well-being, assessing patients' sense of meaning, peace and faith. Items are scored on a five-point Likert scale from 0 (not at all) to 4 (very much), with a total score ranging from 0 to 48, with higher scores indicating higher spiritual wellbeing.
Quality of life, measured by Quality of Life at the End of Life Cancer Scale - Quality of life | Baseline, after 3 months and after 6 months
  The Quality of Life at the End of Life-Cancer Scale (QUAL-EC)is a self- report measure of quality of life in patients near the end of life. It originally consists of five subscales: symptom control, relationship with health care providers, preparation for end of life and life completion. For this study purposes, the symptom control subscale is not included, thus only items 4-17 are used assessing the remaining subscales. Items are scored on a five-point Likert scale ranging from 1 (not at all) to 5 (completely), with a total score ranging from 14 to 70 and higher scores indicating higher quality of life.
Attachment security , measured by ECR-M16 - attachment security | Baseline, after 3 months and after 6 months
  The Experiences in Close Relationships Inventory Modified Short Form Version (ECR-M16), is used in its 16-item self-report form to measure the attachment style (i.e. style in relationships perceived to be important for felt security). The scale yields scores on two dimensions: avoidance and anxiety. Items are scored on a seven-point Likert scale ranging from 1 (disagree) to 7 (agree), with a total sum score ranging from 16 to 56 on each subscale. Higher scores on one or both subscale indicate higher attachment insecurity.
Personal growth measured by PTGI-post-traumatic growth scale | Baseline, after 3 months and after 6 months
  The Posttraumatic Growth Inventory (PTGI) is a 21-item self-report scale which measures positive psychological changes after trauma. It consists of four subscales: new possibilities, appreciation of life, relating to others and spiritual change. Items are scored on a three-point Likert scale ranging from 0 (not at all) to 2 (very much) with a total score ranging from 0 to 42. High scores indicate greater post-traumatic growth.
Communication with partner measured by CCS- communication with partner | Baseline, after 3 months and after 6 months
  The Couple Communication Scale (CCS) is used for participants who are married, common-law, or in a long-term relationship. The CCS is taken from the PREPARE/ENRICH Inventory, of which we used ten items concerning romantic relationship, with each item scored from 1 (strongly disagree) to 5 (strongly agree).
Satisfaction with care, measured by CEQ - satisfaction with care | After 3 and 6 months
  Intervention and control participants complete respectively the Clinical Evaluation Questionnaire (CEQ) [19] - CALM and SPI at 3 and 6-months; a seven-item self-report questionnaire which assesses the level of mastery and insight patients have gained in time and the extent to which therapeutic sessions were perceived as helpful for patients. Experimental group patients' satisfaction will also be qualitatively assessed by inviting participants to share comments in a written form after completing CEQ questionnaire.
Demoralization levels, measured by DS scale - demoralization | Baseline, after 3 months and after 6 months
  The Death and Dying Distress Scale (DADDS) is a 15-item self-report measure assessing specific concerns of advanced cancer patients about end of life, feeling a burden to others and wasted opportunities. It is scored on a six-point Likert scale from 0 (no distress) to 5 (very much distress), with a total score ranging from 0 to 75, a greater score indicating higher death anxiety and distress.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Grassi, M.D., Study Chair — Istituto di Psichiatria. Università degli Studi di Ferrara; Rosangela Caruso, M.D., PhD, Principal Investigator — Istituto di Psichiatria. Università degli Studi di Ferrara
Locations (1):
- Università di Ferrara, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miovic M, Block S. Psychiatric disorders in advanced cancer. Cancer. 2007 Oct 15;110(8):1665-76. doi: 10.1002/cncr.22980. PMID 17847017
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Lloyd-Williams M, Shiels C, Taylor F, Dennis M. Depression--an independent predictor of early death in patients with advanced cancer. J Affect Disord. 2009 Feb;113(1-2):127-32. doi: 10.1016/j.jad.2008.04.002. Epub 2008 Jun 16. PMID 18558439
- [Background] Vehling S, Oechsle K, Koch U, Mehnert A. Receiving palliative treatment moderates the effect of age and gender on demoralization in patients with cancer. PLoS One. 2013;8(3):e59417. doi: 10.1371/journal.pone.0059417. Epub 2013 Mar 15. PMID 23555030
- [Background] Hui D, de la Cruz M, Thorney S, Parsons HA, Delgado-Guay M, Bruera E. The frequency and correlates of spiritual distress among patients with advanced cancer admitted to an acute palliative care unit. Am J Hosp Palliat Care. 2011 Jun;28(4):264-70. doi: 10.1177/1049909110385917. Epub 2010 Nov 7. PMID 21057143
- [Background] Pringle J, Johnston B, Buchanan D. Dignity and patient-centred care for people with palliative care needs in the acute hospital setting: A systematic review. Palliat Med. 2015 Sep;29(8):675-94. doi: 10.1177/0269216315575681. Epub 2015 Mar 23. PMID 25802322
- [Background] Vehling S, Lehmann C, Oechsle K, Bokemeyer C, Krull A, Koch U, Mehnert A. Is advanced cancer associated with demoralization and lower global meaning? The role of tumor stage and physical problems in explaining existential distress in cancer patients. Psychooncology. 2012 Jan;21(1):54-63. doi: 10.1002/pon.1866. Epub 2010 Nov 8. PMID 21061407
- [Background] de Figueiredo J. Diagnosing demoralization in consultation psychiatry. Psychosomatics. 2000 Sep-Oct;41(5):449-50. doi: 10.1176/appi.psy.41.5.449. No abstract available. PMID 11015637
- [Background] Shader RI. Demoralization revisited. J Clin Psychopharmacol. 2005 Aug;25(4):291-2. doi: 10.1097/01.jcp.0000172072.58388.74. No abstract available. PMID 16012269
- [Background] Slavney PR. Diagnosing demoralization in consultation psychiatry. Psychosomatics. 1999 Jul-Aug;40(4):325-9. doi: 10.1016/S0033-3182(99)71227-2. PMID 10402879
- [Background] Robinson S, Kissane DW, Brooker J, Burney S. A systematic review of the demoralization syndrome in individuals with progressive disease and cancer: a decade of research. J Pain Symptom Manage. 2015 Mar;49(3):595-610. doi: 10.1016/j.jpainsymman.2014.07.008. Epub 2014 Aug 15. PMID 25131888
- [Background] Tang PL, Wang HH, Chou FH. A Systematic Review and Meta-Analysis of Demoralization and Depression in Patients With Cancer. Psychosomatics. 2015 Nov-Dec;56(6):634-43. doi: 10.1016/j.psym.2015.06.005. Epub 2015 Jun 19. PMID 26411374
- [Background] Grassi L, Nanni MG. Demoralization syndrome: New insights in psychosocial cancer care. Cancer. 2016 Jul 15;122(14):2130-3. doi: 10.1002/cncr.30022. Epub 2016 May 12. No abstract available. PMID 27171755
- [Background] Faller H, Schuler M, Richard M, Heckl U, Weis J, Kuffner R. Effects of psycho-oncologic interventions on emotional distress and quality of life in adult patients with cancer: systematic review and meta-analysis. J Clin Oncol. 2013 Feb 20;31(6):782-93. doi: 10.1200/JCO.2011.40.8922. Epub 2013 Jan 14. PMID 23319686
- [Background] Walker J, Sawhney A, Hansen CH, Ahmed S, Martin P, Symeonides S, Murray G, Sharpe M. Treatment of depression in adults with cancer: a systematic review of randomized controlled trials. Psychol Med. 2014 Apr;44(5):897-907. doi: 10.1017/S0033291713001372. Epub 2013 Jun 19. PMID 23778105
- [Background] LeMay K, Wilson KG. Treatment of existential distress in life threatening illness: a review of manualized interventions. Clin Psychol Rev. 2008 Mar;28(3):472-93. doi: 10.1016/j.cpr.2007.07.013. Epub 2007 Aug 7. PMID 17804130
- [Background] Nissim R, Freeman E, Lo C, Zimmermann C, Gagliese L, Rydall A, Hales S, Rodin G. Managing Cancer and Living Meaningfully (CALM): a qualitative study of a brief individual psychotherapy for individuals with advanced cancer. Palliat Med. 2012 Jul;26(5):713-21. doi: 10.1177/0269216311425096. Epub 2011 Oct 31. PMID 22042225
- [Background] Lo C, Hales S, Rydall A, Panday T, Chiu A, Malfitano C, Jung J, Li M, Nissim R, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully: study protocol for a randomized controlled trial. Trials. 2015 Sep 3;16:391. doi: 10.1186/s13063-015-0811-1. PMID 26335704
- [Background] Lo C, Hales S, Jung J, Chiu A, Panday T, Rydall A, Nissim R, Malfitano C, Petricone-Westwood D, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): phase 2 trial of a brief individual psychotherapy for patients with advanced cancer. Palliat Med. 2014 Mar;28(3):234-42. doi: 10.1177/0269216313507757. Epub 2013 Oct 29. PMID 24170718
- [Background] Scheffold K, Philipp R, Engelmann D, Schulz-Kindermann F, Rosenberger C, Oechsle K, Harter M, Wegscheider K, Lordick F, Lo C, Hales S, Rodin G, Mehnert A. Efficacy of a brief manualized intervention Managing Cancer and Living Meaningfully (CALM) adapted to German cancer care settings: study protocol for a randomized controlled trial. BMC Cancer. 2015 Aug 19;15:592. doi: 10.1186/s12885-015-1589-y. PMID 26286128
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kissane DW, Wein S, Love A, Lee XQ, Kee PL, Clarke DM. The Demoralization Scale: a report of its development and preliminary validation. J Palliat Care. 2004 Winter;20(4):269-76. PMID 15690829
- [Background] Grassi L, Costantini A, Kissane D, Brunetti S, Caruso R, Piazza G, Marchetti P, Sabato S, Nanni MG. The factor structure and use of the Demoralization Scale (DS-IT) in Italian cancer patients. Psychooncology. 2017 Nov;26(11):1965-1971. doi: 10.1002/pon.4413. Epub 2017 Mar 27. PMID 28263003
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Lo C, Burman D, Swami N, Gagliese L, Rodin G, Zimmermann C. Validation of the QUAL-EC for assessing quality of life in patients with advanced cancer. Eur J Cancer. 2011 Mar;47(4):554-60. doi: 10.1016/j.ejca.2010.10.027. Epub 2010 Dec 1. PMID 21126869
- [Background] Lo C, Hales S, Zimmermann C, Gagliese L, Rydall A, Rodin G. Measuring death-related anxiety in advanced cancer: preliminary psychometrics of the Death and Dying Distress Scale. J Pediatr Hematol Oncol. 2011 Oct;33 Suppl 2:S140-5. doi: 10.1097/MPH.0b013e318230e1fd. PMID 21952572
- [Background] Lo C, Walsh A, Mikulincer M, Gagliese L, Zimmermann C, Rodin G. Measuring attachment security in patients with advanced cancer: psychometric properties of a modified and brief Experiences in Close Relationships scale. Psychooncology. 2009 May;18(5):490-9. doi: 10.1002/pon.1417. PMID 18821528
- [Background] Olson DH, Larson PJ. PREPARE/ENRICH: Customized Version. Life Innovations, Minneapolis. 2008.
- [Background] Vos J. Meaning and existential givens in the lives of cancer patients: A philosophical perspective on psycho-oncology. Palliat Support Care. 2015 Aug;13(4):885-900. doi: 10.1017/S1478951514000790. Epub 2014 Jun 26. PMID 24967611
- [Background] Rodin G, Walsh A, Zimmermann C, Gagliese L, Jones J, Shepherd FA, Moore M, Braun M, Donner A, Mikulincer M. The contribution of attachment security and social support to depressive symptoms in patients with metastatic cancer. Psychooncology. 2007 Dec;16(12):1080-91. doi: 10.1002/pon.1186. PMID 17464942
- [Background] Grassi L, Riba M. Introducing multicultural perspectives in psycho-oncology. In Grassi L., Riba M. (Eds.), Clinical Psycho-Oncology: An International Perspective. Wiley, Chichester, 2012, pp 1-9
- [Background] Grassi L, Caruso R, Nanni M.G.Psycho-oncology and optimal standards of cancer care: developments, multidisciplinary team approach and international guidelines. In Wise T.N., Biondi M., Costantini A. (Eds.), Psycho-Oncology. American Psychiatric Publishing Press, Arlington, VA, 2013, pp 315-339